CLINICAL TRIAL: NCT01308736
Title: Varenicline-Aided Cigarette Reduction in Smokers Not Ready to Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Marc L. Steinberg, Ph.D., Associate Professor, Rutgers University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WS777117
Record Dates: First submitted 2011-01-28; First posted 2011-03-04 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco; nicotine; cigarette smoking
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- varenicline (Active Comparator)
  Interventions: Drug: Varenicline
- placebo pill (Placebo Comparator)
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Varenicline — Participants randomized to receive varenicline will follow the Pfizer recommended dosing schedule (0.5 mg QD on days 1-3, 0.5 mg BID on days 4-7, and 1 mg BID thereafter.
  Arms: varenicline
Drug: Placebo pill — Participants randomized to receive placebo pill will follow the same dosing schedule as those randomized to receive varenicline (1 pill labelled 0.5 mg on days 1-3, pills labelled 0.5 mg BID on days 4-7, and pills labelled 1 mg BID thereafter.
  Arms: placebo pill

SUMMARY:
The investigators will randomize smokers to receive 1) Varenicline + smoking cessation/reduction counseling or 2) Placebo pill + smoking cessation/reduction counseling. Neither the participants nor the research therapists/evaluators will know to which condition (active or placebo pill) the participants have been assigned i.e., a double-blind study). The medication and weekly counseling will occur for 28 days. Participants will complete assessment measures just before the start of treatment (baseline), at the end-of-treatment, at 1-month, 3-month, and at 6-months to determine if there are differences in tobacco use between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Must smoke at least 10 cigarettes per day for past 6-months
* Must have a working cellular or land-line phone

Exclusion Criteria:

* Must not be thinking of quitting in the next 30 days, but be interested in cutting down- Must not regularly (more than 1x/month) use tobacco products other than cigarettes
* Must not be currently receiving tobacco dependence treatment counseling
* Must not currently be taking varenicline, bupropion, nortriptyline, or any nicotine preparations (gum, lozenge, patch, spray, inhaler)
* Must not have positive screen on SCID-I/NP Psychotic Screen
* Must have no contraindications to using varenicline, including pregnancy, as measured by Medical History Form

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc L Steinberg, Ph.D., Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- Division of Addiction Psychiatry, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 73 potential participants provided informed consent and were therefore "Enrolled," however 10 of these did not meet all eligibility criteria as they were completing the baseline measures. We therefore "Started" 63 randomized participants as indicated in the Participant Flow module.
Period: Overall Study
Arm/Group | Varenicline | Placebo Pill
Started | 31 | 32
Completed | 25 | 27
Not Completed | 6 | 5
Not completed — Did not attend a single session | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo Pill | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.03 (10.54) | 44.81 (12.14) | 44.43 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Reduction
Description: 50% reduction in cigarettes per day as compared to baseline. Missing data are assumed to NOT have reduced.
Time Frame: At 6-month follow-up
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo Pill
Number analyzed (Participants) | 31 | 32
participants | 10 | 11

ADVERSE EVENTS:
Arm/Group | Varenicline | Placebo Pill
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 17/31 | 16/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=31) | Placebo Pill (N=32)
Bloating (Gastrointestinal disorders) | 1 | 0
Vivid or Bizarre Dreams (General disorders) | 6 | 4
Nausea (Gastrointestinal disorders) | 9 | 5
Constipation (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 4
Irritability (General disorders) | 2 | 2
Restlessness (General disorders) | 1 | 1
Upset stomach (Gastrointestinal disorders) | 2 | 0
Headache (General disorders) | 1 | 2
Dizzy/light-headed (General disorders) | 3 | 0
Insomnia or fitful sleep (General disorders) | 1 | 3
Sexual dysfunction (General disorders) | 1 | 1
Abdominal cramps (Gastrointestinal disorders) | 1 | 0
Toothache (General disorders) | 1 | 0
Congestion (General disorders) | 2 | 0
Increased depressive symptoms (Psychiatric disorders) | 2 | 2
Fatigue (General disorders) | 2 | 2
Cold/Flu symptoms (General disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Increased appetite (General disorders) | 1 | 0
Blunted affect (Psychiatric disorders) | 0 | 1
Itchy (General disorders) | 0 | 1
Hot flashes (Endocrine disorders) | 0 | 1
Chest twitches (Cardiac disorders) | 0 | 1
Pulled muscle in back (General disorders) | 0 | 1
Gas (Gastrointestinal disorders) | 0 | 2
Strained bowel movement (Gastrointestinal disorders) | 0 | 1
Dry mouth (General disorders) | 0 | 1
Nose bleed (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No